CLINICAL TRIAL: NCT01248858
Title: A Phase I Open-Label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK2126458 and GSK1120212 Combination Therapy in Subjects With Advanced Solid Tumors.
Brief Title: Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of GSK2126458 and GSK1120212 Combination Therapy in Subjects With Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The reason for termination was lack of tolerability and efficacy of the combination treatment
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113794
Record Dates: First submitted 2010-11-18; First posted 2010-11-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — omipalisib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK2126458 and GSK1120212 (Experimental): The first combination schedule that will be tested involves giving both GSK2126458 and GSK1120212 continuously once a day in the morning until the subjects withdraw from the study. Other dosing schedules with both drugs will also be tested and these schedules are described below GSK2126458 will be dosed twice per day (morning and evening) continuously and GSK1120212 will be dosed once a day in the morning on a continuous schedule. Subjects will be treated with both drugs and remain in the study as long as they are benefiting from therapy. Another schedule that will be tested involves giving GSK2126458 twice each day (morning and evening) on an intermittent schedule (4 days of treatment, 10 days rest, then 4 days treatment, 10 days rest). GSK1120212 will be dosed once each day in the morning on a continuous schedule. Subjects will be treated with both drugs as long as they are benefiting from therapy.
  Interventions: Drug: GSK2126458 and GSK1120212

INTERVENTIONS:
Drug: GSK2126458 and GSK1120212 — GSK2126458 and GSK1120212 are experimental treatments for patients with cancer.

SUMMARY:
This is a Phase I, open-label, dose-escalation study to characterize the safety, tolerability, pharmacokinetic profile, pharmacodynamic profile, and clinical activity of the oral PI3K inhibitor GSK2126458 and the oral MEK inhibitor GSK1120212 dosed in combination in subjects with advanced solid tumors. The study will be conducted in 2 parts, a dose escalation phase and a tumor specific cohort expansion.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study to characterize the safety, tolerability, pharmacokinetic profile, pharmacodynamic profile, and clinical activity of the oral PI3K inhibitor GSK2126458 and the oral MEK inhibitor GSK1120212 dosed in combination in subjects with advanced solid tumors. The study will be conducted in 2 parts, a Part 1 dose escalation phase and a Part 2 tumor specific cohort expansion.

A continuous daily dosing schedule will be utilized initially for both investigational products. The frequency and schedule of dosing may be adjusted based on emerging safety, pharmacokinetics, and pharmacodynamics data.

Once a recommended regimen has been characterized in Part 1, it may be further evaluated in Part 2 . More than one regimen (doses and schedules) may be evaluated in Part 2, based on findings in Part 1.

Subjects eligible for enrollment in Part 2 will have solid tumors with genetic profiles that are likely to benefit from a MEK and PI3K pathway inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older at the time of signing the informed consent.
* Confirmed diagnosis of certain molecular types of colorectal , pancreatic, endometrial, ovarian, breast or bladder cancers or melanoma for which there is no approved or curative treatment. Subjects who refuse standard treatment may be included. Physicians should contact the GSK medical monitor for details about the types of tumors that may be treated in this study.
* All prior treatment related toxicities must be CTCAE (Version 4.0) ≤ Grade 1 (except alopecia) at the time of treatment allocation
* Adequate organ system function.
* Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
* Able to swallow and retain orally administered medication
* Subjects with prior Whipple procedure
* Female or male that is willing to take measures to avoid pregnancy in self or a partner, including abstinence, or double barrier method.

Exclusion Criteria:

* Primary malignancy of the CNS or malignancies related to HIV or solid organ transplant. History of known HIV, known Hepatitis B surface antigen or positive Hepatitis C antibody.
* Chemotherapy, extensive radiotherapy, major surgery, anti-neoplastic antibody or targeted therapy or immunotherapy within 28 days (or 42 days for prior nitrosoureas or mitomycin C) prior to the first dose of investigational products.
* Use of an investigational anti-cancer drug within 28 days or five half-lives, whichever is shorter, prior to the first dose of the investigational products.
* Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for retinal vein occlusion or central serous retinopathy, such as: evidence of new optic disc cupping, evidence of new visual field defects or intraocular pressure >21 mm Hg measured by tonography.
* Current use of anticoagulants (e.g., warfarin, heparin) at therapeutic levels within 14 days prior to the first dose of GSK1120212 or GSK2126458. Low dose (prophylactic) low molecular weight heparin and warfarin are permitted drugs.
* Current use of a prohibited medication
* Previously diagnosed with diabetes mellitus (Type 1 or 2) or steroid-induced hyperglycemia.
* Evidence of severe or uncontrolled systemic diseases.
* Any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Brain metastases, unless previously treated brain metastases with surgery, whole brain radiation, or stereotactic radiosurgery and the disease has been confirmed stable (i.e., no increase in lesion size) for at least 8 weeks with two consecutive MRI scans using contrast prior to dosing with investigational product.
* History of acute coronary syndromes coronary angioplasty, or stenting within the past 6 months.
* History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association.
* QTcF interval > or = 470 msecs. History or evidence of current clinically significant uncontrolled arrhythmias. ubjects wtih controlled atrial fibrillation for > 1 month are eligible.
* Treatment refractory hypertension defined as systolic BP > 140 mmHg and/or diastolic BP > 90 mmHg
* Subjects with intra-cardiac defibrillators or permanent pacemakers
* Known cardiac metastases
* Hypersensitivity to study drugs
* Pregnant females or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-12-03 (Actual); Primary Completion 2014-01-30 (Actual); Study Completion 2015-04-23 (Actual)

PRIMARY OUTCOMES:
To characterize the safety of GSK2126458 and GSK1120212 dosed orally in combination through adverse event assessment and changes in safety assessments including laboratory parameters, vital signs, and ECG parameters. | Subjects continue on study until disease progression or consent withdrawn.

SECONDARY OUTCOMES:
To characterize the tolerability of GSK2126458 and GSK1120212 dosed orally in combination through adverse event assessment and changes in safety assessments including laboratory parameters, vital signs, and ECG parameters. | Subjects continue on study until disease progression or consent withdrawn.
To determine the recommended Phase II regimen(s) of GSK2126458 and GSK1120212 dosed orally in combination based on safety, tolerability, PK and PD markers (e.g. changes from baseline in biomarkers of pathway inhibition). | Subjects continue on study until disease progression or consent withdrawn.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (2):
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Nashville, Tennessee
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Milan, Lombardy, Italy

REFERENCES:
- See also: Results for study 113794 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113794?search=study&b'study_ids=113794'#rs